CLINICAL TRIAL: NCT01307098
Title: An Open-Label Multicenter Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SBC-102 in Adult Participants With Liver Dysfunction Due to Lysosomal Acid Lipase Deficiency
Brief Title: Safety, Tolerability and Pharmacokinetics of SBC-102 (Sebelipase Alfa) in Adult Participants With Lysosomal Acid Lipase Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-CL01
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Cholesterol Ester Storage Disease(CESD); Lysosomal Acid Lipase Deficiency; LAL-Deficiency
Keywords: Enzyme Replacement Therapy (ERT); Lysosomal Storage Disease; Late Onset Lysosomal Acid Lipase (LAL) Deficiency; Acid cholesteryl ester hydrolase deficiency, type 2; Acid lipase disease; Cholesterol ester hydrolase deficiency; LAL Deficiency; LIPA Deficiency; Wolman disease
MeSH Terms: conditions — Cholesterol Ester Storage Disease; Wolman Disease; Lysosomal Storage Diseases | interventions — Sebelipase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sebelipase alfa 0.35 mg/kg (Experimental): Cohort 1: Participants were administered once weekly (qw) infusions of 0.35 mg/kg sebelipase alfa.
  Interventions: Drug: Sebelipase alfa 0.35 mg/kg
- Sebelipase alfa 1 mg/kg (Experimental): Cohort 2: Participants were administered qw infusions of 1 mg/kg sebelipase alfa.
  Interventions: Drug: Sebelipase alfa 1 mg/kg
- Sebelipase alfa 3 mg/kg (Experimental): Cohort 3: Participants were administered qw infusions of 3 mg/kg sebelipase alfa.
  Interventions: Drug: Sebelipase alfa 3 mg/kg

INTERVENTIONS:
Drug: Sebelipase alfa 0.35 mg/kg — Sebelipase alfa is a recombinant human lysosomal acid lipase.
  Other Names: Kanuma; SBC-102
  Arms: Sebelipase alfa 0.35 mg/kg
Drug: Sebelipase alfa 1 mg/kg — Sebelipase alfa is a recombinant human lysosomal acid lipase.
  Other Names: Kanuma; SBC-102
  Arms: Sebelipase alfa 1 mg/kg
Drug: Sebelipase alfa 3 mg/kg — Sebelipase alfa is a recombinant human lysosomal acid lipase.
  Other Names: Kanuma; SBC-102
  Arms: Sebelipase alfa 3 mg/kg

SUMMARY:
This was the first clinical study of SBC-102 (sebelipase alfa) for the treatment of Lysosomal Acid Lipase (LAL) Deficiency. It was an open-label dose escalation study in adult participants with liver dysfunction due to LAL Deficiency and was designed to examine 3 doses of sebelipase alfa. The targeted number for this study was 9 evaluable participants.

DETAILED DESCRIPTION:
The study was composed of a screening period, a treatment period, and a post-treatment follow-up period (including an End of Study visit). Participants who successfully completed screening assessments to determine study eligibility were allocated to 3 sequential cohorts (0.35, 1, or 3 milligrams/kilogram [mg/kg]). Within each cohort, one participant was initially dosed and, if sebelipase alfa was deemed safe and well tolerated in this participant (based on at least 24 hours of monitoring), dosing was allowed to be initiated for the remaining participants in the cohort. Initiation of dosing in the next cohort occurred only after all participants in the preceding cohort had been monitored for at least 5 days after the second infusion, without any evidence of significant safety signals, and an independent Safety Committee had reviewed the cumulative safety data and provided their recommendation on the acceptability of beginning dosing in the next cohort.

Cholesteryl Ester Storage Disease (CESD) is the late onset phenotype for LAL Deficiency, a lysosomal storage disorder, which also has an early onset phenotype known as Wolman disease that primarily affects infants. CESD can present in childhood but often goes unrecognized until adulthood when the underlying pathology is advanced. Many of the signs and symptoms are common to participants with other liver conditions.

CESD is an autosomal recessive genetic condition and is characterized by hepatomegaly, persistently abnormal liver function tests and type II hyperlipidemia. Splenomegaly and evidence of mild hypersplenism may affect some participants. Untreated, CESD may lead to fibrosis, cirrhosis, liver failure and death.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥ 18 and ≤ 65 years of age
* Documented decreased LAL activity
* Evidence of liver involvement

Exclusion Criteria:

* Clinically significant concurrent disease, serious inter-current illness, concomitant medications or other extenuating circumstances
* Clinically significant abnormal values on laboratory screening tests, other than liver function or lipid panel tests
* Aspartate aminotransferase and/or alanine aminotransferase persistently elevated > 3x upper limit of normal at screening
* Previous hemopoietic bone marrow or liver transplant
* Current history of alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-04-25 (Actual); Primary Completion 2012-01-06 (Actual); Study Completion 2012-01-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Stanford, California
  - New York, New York
  - Pittsburgh, Pennsylvania
- Prague, Czechia
- Paris, France
- United Kingdom (2):
  - Cambridge
  - Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Balwani M, Breen C, Enns GM, Deegan PB, Honzik T, Jones S, Kane JP, Malinova V, Sharma R, Stock EO, Valayannopoulos V, Wraith JE, Burg J, Eckert S, Schneider E, Quinn AG. Clinical effect and safety profile of recombinant human lysosomal acid lipase in patients with cholesteryl ester storage disease. Hepatology. 2013 Sep;58(3):950-7. doi: 10.1002/hep.26289. Epub 2013 Mar 28. PMID 23348766
- See also: Website — http://alexion.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened for eligibility for enrollment in this study (LAL-CL01). Nine participants met all enrollment criteria and were enrolled and allocated to 1 of 3 cohorts.
Groups:
- Sebelipase Alfa 0.35 mg/kg: Cohort 1: Participants were administered once weekly (qw) infusions of 0.35 milligrams/kilogram (mg/kg) sebelipase alfa.
Period: Overall Study
Arm/Group | Sebelipase Alfa 0.35 mg/kg | Sebelipase Alfa 1 mg/kg | Sebelipase Alfa 3 mg/kg
Started | 3 | 3 | 3
Received at Least 1 Dose of Study Drug | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received any full or partial dose of sebelipase alfa in this study.
Groups:
- Sebelipase Alfa 0.35 mg/kg: Cohort 1: Participants were administered qw infusions of 0.35 mg/kg sebelipase alfa.
- Total: Total of all reporting groups
Arm/Group | Sebelipase Alfa 0.35 mg/kg | Sebelipase Alfa 1 mg/kg | Sebelipase Alfa 3 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 9
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.57) | 35.3 (14.22) | 27.0 (12.17) | 31.6 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 2 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Reporting TEAEs And Infusion-Related Reactions (IRRs)
Description: Safety and tolerability of sebelipase alfa was primarily assessed by monitoring the number of participants reporting treatment-emergent adverse events (TEAEs), including serious adverse events, and infusion-related reactions (IRRs). The number of participants who discontinued from the study due to a TEAE is also presented. An IRR was defined as any adverse event that occurred between the start of the infusion and 4 hours after completion of the infusion and was assessed by the Investigator as at least possibly related to study drug. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Screening up to Day 52
Population: Safety Analysis Set: All participants who received any full or partial dose of sebelipase alfa in this study.
Measure: Number; unit: participants
Arm/Group | Sebelipase Alfa 0.35 mg/kg | Sebelipase Alfa 1 mg/kg | Sebelipase Alfa 3 mg/kg
Number analyzed (Participants) | 3 | 3 | 3
participants
  TEAEs | 1 | 3 | 3
  SAEs | 0 | 0 | 0
  IRRs | 0 | 0 | 0
  TEAEs Leading to Study Discontinuation | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening up to Day 52
Description: Adverse events were obtained through participant reporting or were elicited by specific questioning or examination of the participant.
Arm/Group | Sebelipase Alfa 0.35 mg/kg | Sebelipase Alfa 1 mg/kg | Sebelipase Alfa 3 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sebelipase Alfa 0.35 mg/kg (N=3) | Sebelipase Alfa 1 mg/kg (N=3) | Sebelipase Alfa 3 mg/kg (N=3)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Catheter site related reaction (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/1 | 1/1 | 0/1 — Affects only female participants
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes